CLINICAL TRIAL: NCT02174484
Title: Pacemaker Remote Electrogram Monitoring Study (PREMS)
Brief Title: Assessment of Intracardiac Electrograms Transmitted by Home Monitoring for the Remote Follow-up of Pacemaker (PREMS)
Acronym: PREMS
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HS057
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Bradycardia
Keywords: Pacemaker; Remote monitoring; Remote follow-up; Home monitoring; Periodic IEGM; Intracardiac electrogram
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker recipients: Patients implanted with a single or dual pacemaker and with Home-Monitoring system activated and periodic IEGM activated

SUMMARY:
The purpose of the PREMS study is to evaluate the capability of the periodic IEGM feature (intracardiac electrogram) to provide more extensive remote information about cardiac rhythm, sensing and capture, and thus to detect anomalies that may deserve a clinical action.

PREMS is a non-interventional, prospective, and multicenter study. The primary objective is to assess the added clinical value of periodic IEGMs, based on the rate of patients with a rhythm or sensing/pacing anomaly detected on the first IEGM transmitted by Home Monitoring (HM) and non detectable so obvious on the other parameter set offered for the remote follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with a single or dual chamber PM within the last 3 months
* Home-Monitoring activated and functional
* Periodic IEGM "ON" and programmed at 30 days intervals
* Patient willing and able to comply with the protocol and who has provided written informed consent about HM
* Patient whose medical situation is stable

Exclusion Criteria:

* Age < 18 years
* Patient unable to handle the Cardio messenger correctly
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted with a single or dual chamber pacemaker and with the Biotronik Home-Monitoring® system activated
Sampling Method: Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Added clinical value of periodic IEGM | 1 month
  The main objective of the study is to evaluate the added clinical value of periodic IEGMs for the remote follow-up of PM, compared to other HM data offered by the remote follow-up.
  Primary endpoint:
  Rate of patients with at least one rhythm or sensing/pacing anomaly detected on the periodic IEGM, and non detectable on the other HM data. The anomalies are defined as an arrhythmia (extrasystole, atrial fibrillation or flutter), loss of sensing, oversensing or loss of capture.

SECONDARY OUTCOMES:
Planned corrective action | 1 month
  Rate of detected anomalies triggering a planned corrective action
Added clinical value of the remote follow-up | 1 month
  Rate of anomalies that can be identified based on remote data other than the periodic IEGM and comparison with the previous event notifications
Type of detected anomalies | 1 month
  The types of anomalies detected on the periodic IEGM or/and on the other HM data will be evaluated separately (arrhythmia, loss of capture, loss of sensing, oversensing)
Capability of periodic IEGM to fulfil the guidelines requirements | 1 month
  The periodic IEGMs transmitted by HM are designed in accordance with ACC/AHA/HRS guidelines. Indeed, guidelines for a PM follow-up require to determine the current intrinsic rhythm, but also to check the appropriate sensing and capture. The periodic IEGM could remotely provide the same information than an in-office follow-up. So, the capability of periodic IEGM to fulfil the requirements for PM follow-up by ACC/AHA/HRS guidelines will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Lazarus, MD, Principal Investigator — Clinique Ambroise Paré, Neuilly sur Seine, France
Locations (49):
- France (49):
  - Clinique Axium, Aix-en-Provence
  - Clinique de l'Anjou, Angers
  - CH d'Annecy, Annecy
  - CH Annonay, Annonay
  - CH d'Antibes, Antibes
  - CH d'Aurillac, Aurillac
  - CH de Bastia, Bastia
  - Clinique Saint Vincent, Besançon
  - CH de Blois, Blois
  - Cabinet de Cardiologie, Bordeaux
  - Polyclinique Nord Aquitaine, Bordeaux
  - CH Pierre Oudot, Bourgoin
  - CH des Broussailles, Cannes
  - CH de Castres, Castres
  - Polyclinique Sevigné, Cesson-Sévigné
  - CH de Chambéry, Chambéry
  - Hôpital Privé Paul d'Egine, Champigny-sur-Marne
  - CH de Chartres, Chartres
  - Clinique Bon Secours, Châtellerault
  - Polyclinique du Parc, Cholet
  - Clinique des Dômes, Clermont-Ferrand
  - CH de Douarnenez, Douarnenez
  - Clinique du Mousseau, Évry
  - Clinique de la Marche, Guéret
  - Cabinet de cardiologie, Le Puy-en-Velay
  - CHG de Longjumeau, Longjumeau
  - CH St Luc St Joseph, Lyon
  - Clinique Clairval, Marseille
  - CH Montbrison, Montbrison
  - CH de Nevers, Nevers
  - Cabinet Descartes, Niort
  - CH de Niort, Niort
  - CH Léon Binet, Provins
  - Polyclinique Saint Laurent, Rennes
  - CH de Roanne, Roanne
  - CHU Hôpital Charles Nicolle, Rouen
  - CH Val d'Ariège, Saint Jean de Verge
  - Clinique de Saint Georges de Didonnes, Saint-Georges-de-Didonne
  - Clinique Belledonne, Saint-Martin-d'Hères
  - CH de Saint Malo, St-Malo
  - Hôpitaux du Léman, Thonon-les-Bains
  - HIA Saint Anne, Toulon
  - Hôpital Sainte Musse CHI, Toulon
  - HPOP, Trappes
  - CH de Valence, Valence
  - Cabinet de cardiologie, Valognes
  - CH André Mignot, Versailles
  - CH Paul Morel, Vesoul
  - CHG Villefranche, Villefranche-sur-Saône